CLINICAL TRIAL: NCT04957511
Title: Pilot Feasibility Study of the Interplay Between the Host Gut Microbiome and Efficacy of Treatment for Advanced or Recurrent Gynecological Cancer Patients Receiving Immunotherapy
Brief Title: Gut Microbiome and Treatment for Gynecological Cancer Patients Receiving Immunotherapy
Status: Recruiting | Type: Observational
Sponsor: Viome (Industry)
Collaborators: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: V235
Record Dates: First submitted 2021-06-10; First posted 2021-07-12 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Gynecologic Cancer; Immunotherapy; Gut Microbiome
Keywords: Biome; Microbiome; Gastrointestinal; Immune check point inhibitors; Nutrition; Diet; Viome; ICI; ICIs; RNAseq; Anti-tumor immunity; Cancer; Gynecology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Only RNA molecules are sequenced, while DNA is degraded. The AdventHealth Research Laboratory will process the de-identified blood samples and store; Plasma, Serum and Buffy Coat for future analysis. The Advent Health Research Laboratory will store these samples in the biorepository, inventory and chain of custody will be managed by the STARLIMS program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
30 participants with advanced or recurrent gynecological cancer from are enrolled for this study. Eligible participants then provide fecal specimen, blood, vaginal swab, oral mucosal swab and receive food dietary recommendation. Additional samples are collected for results analysis.

DETAILED DESCRIPTION:
30 patients diagnosed with advanced or recurrent gynecological cancer who plan to receive immunotherapy treatment with a checkpoint inhibitor at AHMG AdventHealth Orlando Gynecological Oncology Group are recruited. Patients will be recruited 1-2 weeks prior to the beginning of treatment and appropriate informed consent will be obtained. Fecal samples; blood; saliva and vaginal swab samples will be collected among participants prior to their first treatment, after four doses of immunotherapy, and again at the completion of immunotherapy (follow-up). These 4 biomarker samples will undergo metatranscriptomic analysis, also known as RNAseq, method of sample analysis. Only RNA molecules are sequenced, while DNA is degraded. for bacterial community analysis. These findings will help to design a future study to examine the role of the gut microbiome in antitumor immunity and its effect on immune checkpoint inhibitor therapy for advanced or recurrent gynecological cancer. NHANES Food Frequency Questionnaire will be collected prior to participants' first treatments.

The short-term goals of this pilot study are to obtain preliminary data on the gut bacterial microbiome of patients with advanced or recurrent gynecological cancer. The long-term goals of this study is to begin to understand how the gut microbiome changes within an individual patient undergoing immunotherapy, to gut microbiome differs among patients undergoing immunotherapy, and to examine whether the gut microbiome is associated with the response to cancer immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult females > 18 years old
* Advanced or recurrent gynecological cancer patients from AHMG Advent Health Orlando Gynecologic Oncology Group
* Patients for whom an immunotherapy regimen has been ordered

Exclusion Criteria:

* Patients unable to provide fecal specimens at three time points
* Patients unable to read or understand informed consent
* Taking medications that may affect gut microbiome:

  * Proton pump inhibitors (PPIs)
  * Metformin
  * Antibiotics
  * Laxatives
* Patients who are receiving investigational agent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult females >18 years old
Study Population: Advanced or recurrent gynecological cancer patients receiving immunotherapy from AHMG Advent Health Orlando Gynecologic Oncology Group
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Microbiome change through analysis of biological samples (fecal specimen, blood, vaginal swab, oral mucosal swab). | ~2 years
  Changes are measured between the genetic microbiome signatures of advanced or recurrent gynecological cancer patients who are receiving immune checkpoint inhibitors.

CONTACTS AND LOCATIONS:
Overall Officials: Momchilo Vuyisich, PhD, Principal Investigator — Viome Life Sciences
Locations (1):
- AdventHealth Cancer Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided